CLINICAL TRIAL: NCT01585350
Title: A Multipeptide Vaccine Plus Toll-Like Receptor Agonists in Melanoma Patients, With Evaluation of the Injection Site Microenvironment
Brief Title: A Multipeptide Vaccine Plus Toll-Like Receptor Agonists in Melanoma Patients
Acronym: MEL58
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: University of Virginia (Other); National Cancer Institute (NCI) (NIH); Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15781
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma
Keywords: melanoma; peptide vaccine; polyICLC; lipopolysaccharide (LPS); immunotherapy
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Vaccines will be administered subcutaneously, intradermally or transdermally in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: MELITAC 12.1 + Montanide ISA-51 + lipopolysaccharide (LPS)
- Cohort 2 (Experimental): Vaccines will be administered subcutaneously, intradermally or transdermally in one skin location that is rotated to different sites on an extremity clinically uninvolved with melanoma.
  Vaccines will be administered on days 1, 8, 15, 36, 57, and 78.
  Interventions: Biological: MELITAC 12.1 + Montanide ISA-51 + polyICLC

INTERVENTIONS:
Biological: MELITAC 12.1 + Montanide ISA-51 + lipopolysaccharide (LPS) — Cohort 1 will be divided into three sub-groups and will receive:
  * Group 1a: MELITAC 12.1 + lipopolysaccharide (LPS)
  * Group 1b: MELITAC 12.1 + lipopolysaccharide (LPS) + Montanide adjuvant with vaccination #1
  * Group 1c: MELITAC 12.1 + lipopolysaccharide (LPS) adjuvant + Montanide adjuvant with all vaccinations
  Arms: Cohort 1
Biological: MELITAC 12.1 + Montanide ISA-51 + polyICLC — Cohort 2 will be divided into three sub-groups and will receive:
  * Group 2a: MELITAC 12.1 + polyICLC adjuvant
  * Group 2b: MELITAC 12.1 + polyICLC adjuvant + Montanide adjuvant with vaccination #1
  * Group 2c: MELITAC 12.1 + polyICLC adjuvant + Montanide adjuvant with all vaccinations
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to learn the effects an experimental vaccine (MELITAC 12.1) combined with other substances called lipopolysaccharide (LPS; endotoxin), polyICLC, and Montanide ISA-51. The LPS, polyICLC, and Montanide ISA-51 are included with the vaccine to test whether they have an effect on the MELITAC 12.1 vaccine. The study will also look at whether the experimental vaccine and these drugs cause any changes to the immune system.

DETAILED DESCRIPTION:
Goals:

1. To determine the safety of intradermal and subcutaneous injection of lipopolysaccharide (LPS) as a vaccine adjuvant with a multipeptide vaccine.
2. To obtain preliminary data on whether administration of a multipeptide vaccine plus each of 2 TLR agonists is immunogenic with or without Incomplete Freund's Adjuvant (IFA)
3. To obtain preliminary data on whether addition of either of 2 toll-like receptor (TLR) agonists improve the persistence of circulating CD8+ T cell responses to vaccination with a multipeptide vaccine.
4. To determine the local and systemic toxicities of administration of a multipeptide vaccine with each of 2 TLR agonists, and with or without incomplete Freund's adjuvant.
5. To determine the cytokine and chemokine profile of the vaccine-site microenvironment week 1 after injection of a multipeptide vaccine and each of 2 TLR agonists, with or without IFA.
6. To obtain preliminary data on T cell activation status and apoptosis in the vaccine site microenvironment (VSME) as a function of vaccine adjuvant.
7. To assess whether circulating CD8 T cells induced by vaccination express different homing receptor profiles (CLA, CXCR3, α4β1 integrin, α4β7 integrin).
8. To evaluate dendritic cell activation and function in sentinel immunized nodes draining the site of vaccination, for production of IDO, arginase, IL10, IL12.
9. To characterize MyD88 expression in dendritic cells infiltrating vaccination sites.
10. To identify regulatory processes in the vaccination site.

Design: This is an open-label, randomized, pilot study of cellular and molecular events at the cutaneous site of immunization with a multipeptide vaccine. This and related peptide vaccines have been associated with immunologic efficacy in a majority of participants and have been associated with clinical tumor regressions in some participants. The maximum number of participants accrued will be 51.

Endpoints:

Primary:

* Safety, with measures of adverse events, locally and systemically
* CD8+ and CD4+ peptide-reactive T cell responses among lymphocytes in the peripheral blood and in sentinel immunized nodes (SIN)

Secondary:

* Toll-like receptor signaling in the replicate immunization site
* CCR and integrin expression on vaccine induced T cells in the peripheral blood and at the replicate immunization site
* Th1, Th2, and Th17 profiles of T cells in the vaccination site and SIN as measured by cytokine expression (IFNγ, IL-2, TNFα, IL-4, IL-5, IL-10, IL-17, IL-23), and nuclear expression of transcription factors (T-bet, GATA3, RORγt) by immunohistochemistry.
* Chemokines CXCL9, 10, and 11; CCL19, CCL21, CXCL12, CXCL13 in the vaccine site microenvironment.
* Markers of activation, regulation, and apoptosis on CD4 and CD8 T cells in the vaccine site and SIN: CD69, Ki67, FoxP3, and TUNEL staining.
* Homing receptors expressed by antigen-reactive (tetramer-positive) T cells induced by vaccination, in the circulation and SIN.
* MyD88 expression in the VSME and SIN
* Regulatory processes in the immunization site and SIN

  * Regulatory T cells (CD4+CD25hi FoxP3+)
  * Myeloid suppressor cells
  * Indole-amine dioxygenase
  * PD-1, B7-H1
  * IL-10 and IL-12 expression by dendritic cells (DC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven melanoma that meets one of the following two criteria:

  * Stage IIB-IV melanoma rendered clinically free of disease by surgery, other therapy, or spontaneous remission within 6 months prior to registration.
  * Stage III or IV melanoma with disease. Patients may be eligible if there are definite or equivocal findings of persistent or metastatic disease as long as those findings do not meet RECIST criteria for measurable disease.
* Patients with brain metastases may be eligible if all of the following are true:

  * The total number of brain metastases ever is less than or equal to 3.
  * The brain metastases have been completely removed by surgery or have been treated completely by stereotactic radiotherapy. Stereotactic radiotherapy, such as gamma knife, can be used up to 1 week prior to study entry.
  * There has been no evident growth of any brain metastasis since treatment.
  * No treated brain metastasis is greater than 2 cm in diameter at the time of protocol entry.
* Patients must have at least two intact axillary and/or inguinal lymph node basins.
* All patients must have:

  * ECOG performance status of 0 or 1.
  * Ability and willingness to give informed consent.
* Laboratory parameters as follows:

  * HLA-A1, A2, A3, -A11, or -A31
  * ANC > 1000/mm3
  * Platelets > 100,000/mm3
  * Hgb ≥ 9 g/dL
  * AST and ALT ≤ 2.5 x upper limits of normal (ULN)
  * Bilirubin ≤ 2.5 x ULN
  * Alkaline Phosphatase ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN
  * HIV negative
  * Hepatitis C negative
  * HGBA1C level of < 7%

Exclusion Criteria:

* Patients who have had brain metastases, unless they meet inclusion criteria
* Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, or other experimental therapy, or who have received this therapy within the preceding 4 weeks. Gamma knife or stereotactic radiosurgery may be administered within the prior 4 weeks, but must not be administered less than one week prior to study enrollment. Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks.
* Patients with clinically detectable melanoma deemed likely by the investigator to require intervention during the first 12 weeks of the study that would require premature discontinuation.
* Patients with known or suspected allergies to any component of the vaccine.
* Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded:

  * Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents and topical steroids
  * Allergy desensitization injections.
  * Systemic corticosteroids, administered parenterally or orally. Inhaled steroids (e.g. Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex®).
  * Any growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
  * Interferon therapy.
  * Interleukin-2 or other interleukins.
  * Toll-like receptor agonists, including imiquimod or resiquimod.
* Prior melanoma vaccinations may be an exclusion criterion in some circumstances:

  * Patients who have recurred or progressed either after or during administration of a melanoma vaccine may be eligible to enroll 12 weeks following their last vaccination.
  * Patients may have been vaccinated previously with peptide vaccines (except that they may not have been vaccinated with peptides included in MELITAC 12.1 or MELITAC 12.6)
  * Patients may have been vaccinated with protein, DNA, or cell-based vaccines that include the proteins from which these peptides are derived.
* Other investigational drugs or investigational therapy if the patient is currently taking those drugs/therapy, or if they have received the drugs/therapy within 1 month.
* Pregnancy or the possibility of becoming pregnant during vaccine administration. Women must also not be breast feeding.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified as having Class III or IV heart disease according to the New York Heart Association
* Body weight < 110 lbs
* No active or prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. The following will not be exclusionary:

  * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without associated symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring NSAID medications or no medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety, with measures of adverse events, locally and systemically | over 6 months
CD8+ and CD4+ peptide-reactive T cell responses among lymphocytes in the peripheral blood and in sentinel immunized nodes (SIN) | over 6 months

SECONDARY OUTCOMES:
Toll-like receptor signaling in the replicate immunization site | over 6 months
CCR and integrin expression on vaccine induced T cells in the peripheral blood and at the replicate immunization site | over 6 months
Th1, Th2, and Th17 profiles of T cells in the vaccination site and SIN as measured by cytokine expression (IFNγ, IL-2, TNFα, IL-4, IL-5, IL-10, IL-17, IL-23), and nuclear expression of transcription factors (T-bet, GATA3, RORγt) by immunohistochemistry. | over 6 months
Chemokines CXCL9, 10, and 11; CCL19, CCL21, CXCL12, CXCL13 in the vaccine site microenvironment | over 6 months
Markers of activation, regulation, and apoptosis on CD4 and CD8 T cells in the vaccine site and SIN: CD69, Ki67, FoxP3, and TUNEL staining | over 6 months
Homing receptors expressed by antigen-reactive (tetramer-positive) T cells induced by vaccination, in the circulation and SIN | over 6 months
MyD88 expression in the VSME and SIN | over 6 months
Regulatory processes in the immunization site and SIN | over 6 months
  * Regulatory T cells (CD4+CD25hi FoxP3+)
  * Myeloid suppressor cells
  * Indole-amine dioxygenase
  * PD-1, B7-H1
  * IL-10 and IL-12 expression by dendritic cells (DC)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Pollack KE, Meneveau MO, Melssen MM, Lynch KT, Koeppel AF, Young SJ, Turner S, Kumar P, Sol-Church K, Mauldin IS, Slingluff CL Jr. Incomplete Freund's adjuvant reduces arginase and enhances Th1 dominance, TLR signaling and CD40 ligand expression in the vaccine site microenvironment. J Immunother Cancer. 2020 Apr;8(1):e000544. doi: 10.1136/jitc-2020-000544. PMID 32350119
- [Derived] Melssen MM, Petroni GR, Chianese-Bullock KA, Wages NA, Grosh WW, Varhegyi N, Smolkin ME, Smith KT, Galeassi NV, Deacon DH, Gaughan EM, Slingluff CL Jr. A multipeptide vaccine plus toll-like receptor agonists LPS or polyICLC in combination with incomplete Freund's adjuvant in melanoma patients. J Immunother Cancer. 2019 Jun 27;7(1):163. doi: 10.1186/s40425-019-0625-x. PMID 31248461